CLINICAL TRIAL: NCT00392262
Title: An Multicenter Study to Evaluate the Efficacy and Tolerability of a 4-week Therapy With the Combination of Valsartan 160mg + Amlodipine 5mg in Hypertensive Patients Not Adequately Responding to 4-week Treatment With Amlo 5mg or Felodipine 5mg in Monotherapy
Brief Title: A Study to Evaluate the Combination of Valsartan + Amlodipine in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489ADE03
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Moderate essential hypertension (WHO grade II)
MeSH Terms: conditions — Hypertension; Lymphoma, Follicular | interventions — Amlodipine, Valsartan Drug Combination

INTERVENTIONS:
Drug: valsartan + amlodipine

SUMMARY:
The purpose of this study is to evaluate the efficacy of valsartan plus amlodipine in hypertensive patients not responding to treatment with amlodipine or felodipine alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients (18 years)
2. Patients with moderate essential hypertension (untreated must have MSSBP ≥160 and <180 mmHg at Visit 1, treated must have MSSBP <180 mmHg at Visit 1) (WHO grade II)

Exclusion Criteria:

1. Severe hypertension(MSDBP ≥110 mmHg or MSSBP ≥ 180 mmHg)
2. Pregnant or nursing women
3. Treated hypertensive patients with controlled hypertension under current therapy (diastolic BP < 90 mmHg and systolic BP < 140 mmHg)
4. A history of cardiovascular disease, including angina pectoris, myocardial infarction, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, transient ischemic attack, stroke, and heart failure NYHA II - IV

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2006-08; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To investigate whether 4 weeks treatment with valsartan 160mg + amlo 5mg provide an add'l mean sitting systolic blood pressure reduction in patients not adequately responding to 4 weeks treatment with amlo 5mg or felodipine 5mg

SECONDARY OUTCOMES:
Mean sitting diastolic blood pressure (analogously & explorative)
Normalization (analogously & explorative)
Responder rate. (analogously & explorative)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis +41 61 324 1111, Study Director — Novartis
Locations (2):
- Investigative Centers, Germany
- Novartis, Basel, Switzerland

REFERENCES:
- [Result] Brachmann J, Ansari A, Mahla G, Handrock R, Klebs S. Effective and safe reduction of blood pressure with the combination of amlodipine 5 mg and valsartan 160 mg in hypertensive patients not controlled by calcium channel blocker monotherapy. Adv Ther. 2008 May;25(5):399-411. doi: 10.1007/s12325-008-0054-6. PMID 18465097